CLINICAL TRIAL: NCT00229125
Title: Gabapentin Vs. Lorazepam in Alcohol Withdrawal
Brief Title: Comparing the Treatment of Alcohol Withdrawal Syndrome Using Gabapentin Versus Lorazepam
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIAAAMAL10761-b; NIH P-50-AA010761
Record Dates: First submitted 2005-09-27; First posted 2005-09-29 (Estimated); Last update posted 2005-09-29 (Estimated); Status verified 2005-09

CONDITIONS: Alcohol Withdrawal Syndrome(AWS)
Keywords: Alcohol Withdrawal Syndrome; CIWA-Ar; Acoustic Startle Procedure; Rebound Effect
MeSH Terms: interventions — Gabapentin; Lorazepam

INTERVENTIONS:
Drug: Gabapentin
Drug: Lorazepam

SUMMARY:
The purpose of this study was to evaluate if the medication Gabapentin, which is not approved for the treatment of alcohol withdrawal, is effective in the treatment of alcohol withdrawal syndrome compared to treatment with Lorazepam.

DETAILED DESCRIPTION:
In the current protocol we evaluated a newer generation anticonvulsant agent, gabapentin. Gabapentin does not significantly interact with alcohol or other medications, has no abuse potential, and is excreted by the kidneys and not the liver .

The primary aim of the present application was to evaluate the efficacy of gabapentin in comparison to lorazepam (as a benzodiazepine gold standard) for the acute outpatient treatment of alcohol withdrawal (AW). In addition, evaluation of the lorazepam "rebound" effects observed during the current funding period will be replicated and compared with the response to gabapentin. Also, the acoustic startle response was used to evaluate the neurobiological effects of the medications on underlying AW-related CNS excitation, both during and immediately after AW. In addition, the effect of a history of multiple detoxifications on parameters such as withdrawal symptoms, CNS excitability, relapse to alcohol use, craving for alcohol, and response to medication treatment was explored.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be between 21-70 years of age (both genders will be recruited).
* Subjects must meet DSM-IV criteria for alcohol dependence and uncomplicated alcohol withdrawal syndrome.
* Subjects must have a mini-mental state score above 26.
* Subjects must be medically stable (not likely to require hospitalization for medical complications within 10 days).
* Subjects must have a minimum score on the Clinical Institute Withdrawal - - Assessment for Alcohol-Revised (CIWA-Ar) of 10 within 24 hours of initial assessment.
* Subjects must be medically acceptable for study treatment. Considerations include no past or present physical disorder that is likely to deteriorate during participation. No ECG abnormality which would likely worsen during participation and no clinical laboratory abnormality that would also suggest deterioration during treatment.
* Subjects must exhibit vital signs within the following range: a three-minute sitting blood pressure in the range of 90-200 mmHg systolic, 60-120 mmHg diastolic and ventricular rates between 56 and 140 beats per minute.
* Subjects must be suitable for treatment with oral medications.
* Subjects must be able to read, write, and speak English.
* Subjects must have a negative urine drug screen for benzodiazepines or other sedative-hypnotics, opiates, and stimulants at baseline.

Exclusion Criteria:

* Subjects with current (past month) DSM-IV diagnosis of any other substance dependence syndrome other than alcohol dependence (excluding nicotine, caffeine, cannabis and cocaine dependence).
* Use of pharmacological agents within a five half-life period that are known to lower the seizure threshold or augment or decrease the alcohol withdrawal syndrome (e.g.,tricyclic antidepressants, anticonvulsants, neuroleptics, benzodiazepines, some centrally-acting antihypertensives such as beta-blockers, alpha-adrenergic agonists, and calcium channel antagonists, wellbutrin, buspar, any sedative-hypnotics and opiates).
* Subjects with a history of idiopathic epilepsy.
* Subjects with diagnosis of schizophrenia, bipolar disorder or dementia.
* Subjects with liver function tests (AST or ALT) 4 times higher than normal. Serum levels will be drawn upon admission to study and study medications terminated if necessary.
* History of hepatic encephalopathy, jaundice, ascites, insulin dependent diabetes, or renal disease.
* Females who are pregnant (as determined by a pregnancy test) or nursing.
* Subjects with known sensitivity or previous adverse reaction to gabapentin, lorazepam, or other benzodiazepines.
* History of severe GI disease which might render absorption of the medication difficult or produce medical instability of the patient during detoxification which would include active peptic ulcer disease, ulcerative colitis, regional colitis, or evidence by history or physical exam of GI bleeding.
* Subjects who decline or who are not competent to give informed consent.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160
Dates: Start 2001-07; Study Completion 2005-09

PRIMARY OUTCOMES:
Clinical Institute Withdrawal Assessment for Alcohol (CIWA-Ar).
Timeline Followback (TLFB) of drinking behaviors.

SECONDARY OUTCOMES:
Lower startle reflex magnitudes as an index of CNS excitability or arousal.
Lower anxiety (Zung Anxiety Scale) and depression (Beck Depression.
Inventory) scores.
Subjective reports of sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Robert J. Malcolm, MD, Principal Investigator — Medical University of South Carolina; Carrie Randall, PhD, Study Director — Medical University of South Carolina, Center for Drug and Alcohol Programs
Locations (1):
- Medical University of South Carolina - Center for Drug and Alcohol Programs, Charleston, South Carolina, United States